CLINICAL TRIAL: NCT04794452
Title: Dental Plaque Removal Evaluation and Comparison of Kid's Battery-Operated Toothbrush
Brief Title: Dental Plaque Removal Evaluation and Comparison of Kid's Battery-Operated Toothbrush and Manual Toothbrush
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Church & Dwight Company, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: ST-20-U82
Record Dates: First submitted 2021-02-14; First posted 2021-03-12 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Plaque, Dental
MeSH Terms: conditions — Dental Plaque

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Battery operated toothbrush (Active Comparator): battery operated toothbrush
  Interventions: Device: Battery operated toothbrush
- Manual toothbrush (Active Comparator): Manual toothbrush
  Interventions: Device: Manual toothbrush

INTERVENTIONS:
Device: Battery operated toothbrush — Device on plaque removal efficacy
  Arms: Battery operated toothbrush
Device: Manual toothbrush — Device on plaque removal efficacy
  Arms: Manual toothbrush

SUMMARY:
To evaluate and compare the plaque removal efficacy of a children's battery-powered toothbrush and a children's manual toothbrush following a single brushing.

DETAILED DESCRIPTION:
This is a single use, examiner blinded, randomized, two-period, cross-over, IRB-approved research study evaluating the single-use plaque removal efficacy of a new children's battery-operated toothbrush and a marketed children's manual toothbrush. This study will accept up to 60 juvenile subjects, 5-8 years of age, in anticipation that 50 subjects will complete the study. Qualified subjects with sufficient plaque, according to Rustogi Modified Navy Plaque Index (RMNPI) will be randomly assigned to one of two sequence treatment groups.

After the pre-brushing plaque evaluation at each of the evaluation visits, subjects will brush with the assigned toothbrush and toothpaste provided for timed brushing under supervision, in front of mirror.

ELIGIBILITY:
Inclusion Criteria:

1. 5 to 8 years
2. Be a regular manual toothbrush user.

Exclusion Criteria:

1. Have any physical limitations or restrictions which might preclude normal tooth brushing.
2. Have evidence of poor oral hygiene or rampant dental caries or presence of extrinsic stain or calculus deposits that may interfere with plaque assessments.
3. Have fixed or removable orthodontic appliances.

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2020-11-23 (Actual); Primary Completion 2020-12-11 (Actual); Study Completion 2020-12-11 (Actual)

PRIMARY OUTCOMES:
Within-Treatment Whole-Mouth Differences (vs Baseline) - Plaque removal | up to 2 weeks
  Mean Change from baseline (pre-brushing to post-brushing) in plaque score after single supervised use based on all surfaces of the whole mouth measured.

CONTACTS AND LOCATIONS:
Locations (1):
- All Sum Research Center Ltd., Mississauga, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No